CLINICAL TRIAL: NCT06197724
Title: Magnetocardiography as an Innovative Diagnostic Tool for Early and Accurate Identification of Myocardial Ischemia in Suspected NSTE-ACS Patients
Brief Title: MCG for Identification of Myocardial Ischemia in Suspected NSTE-ACS Patients
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Linyi People's Hospital (Other); Weifang People's Hospital (Other); Jining First People's Hospital (Other); Weihai Central Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); First People's Hospital of Hangzhou (Other); Chongqing Emergency Medical Center (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Qianfoshan Hospital (Other); Heze Municipal Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: MCG-NSTEACS
Record Dates: First submitted 2023-12-11; First posted 2024-01-09 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Non ST Segment Elevation Acute Coronary Syndrome
MeSH Terms: interventions — Magnetocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training and testing cohort
  Interventions: Device: Magnetocardiography
- External validation cohort
  Interventions: Device: Magnetocardiography

INTERVENTIONS:
Device: Magnetocardiography — Magnetocardiography

SUMMARY:
The goal of this multi-center observational study is to learn about the effectiveness of magnetocardiography in rapid and accurate identification of ischemia in patients with suspected NSTE-ACS.

DETAILED DESCRIPTION:
Rapid and accurate Identification of ischemia in patients with chest pain suspected of non-ST-elevation-acute coronary syndrome (NSTE-ACS) is of great clinical significance for timely and effective treatment. Magnetocardiography based on spin-exchange relaxation-free (SERF) principle can detect the weak magnetic field generated by the heart sensitively, which do not need ultra-low temperature cooling. Magnetic signal does not decay through the skin and tissues as electricity does, hence magnetocardiogram (MCG) contains more information of diagnostic value of ischemia. The aim of this observational study is to optimize and validate MCG models as a fast and accurate strategy for detecting coronary ischemia, as a shortage of blood supply to myocardium, in patients who suffer from chest pain, and compare to routine diagnostic means.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Patients with symptoms of myocardial ischemia such as angina who are suspected to NSTE-ACS and proposed to undergo CAG or coronary CTA;
3. Signed informed consent.

Exclusion Criteria:

1. Patients with ST-elevation myocardial infarction (STEMI);
2. Patients with Non-ischemic dilated cardiomyopathy, or hypertrophic cardiomyopathy, or moderate or severe valvular disease;
3. Patients with Hemodynamic instability (systolic blood pressure<90 mmHg, or who requires vasoactive drugs), or patients with tachyarrhythmia, Ⅱ degree atrioventricular block and above that have not returned to normal;
4. Patients who have severe renal abnormality with eGFR <30 ml/min, or patients who are on dialysis;
5. Patients with malignant tumors with predicted survival of less than 1 year;
6. Pregnant or breastfeeding women;
7. Patients who are unable to enter the MCG device, who are unable to perform MCG examination due to interference from metal implants or other reasons, or who are deemed by the investigators to be unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chest pain patients with suspected NSTE-ACS
Sampling Method: Non-Probability Sample
Enrollment: 14090 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of MCG to detect coronary ischemia in patients with suspected NSTE-ACS | from the date of enrollment until the date of discharge, up to 30 days
  the sensitivity and specificity of MCG to detect coronary ischemia (defined as stenosis ≥ 90% or fractional flow reserve ≤0.8）

SECONDARY OUTCOMES:
Efficacy of MCG in identifying coronary ischemia in patients with normal ECG. | from the date of enrollment until the date of discharge, up to 30 days
  A normal ECG is determined by two cardiologists with over five years of working experience. If there is any objection, the decision shall be made by a third cardiologist of the same qualifications or above. Sensitivity, specificity, and area under ROC curve (AUC) are performed for assessing the efficacy.
The time saved by using MCG in the detection of NSTEMI compared to troponin | from the date of enrollment until the date of discharge, up to 30 days
  The time for the detection of NSTEMI is from the timepoint of first medical contact to the timepoint of MCG report showing ischemia or the first report of troponin that over the 99th percentile of the Upper reference limit (URL).
Efficacy of MCG in evaluating the severity of coronary lesions. | from the date of enrollment until the date of discharge, up to 30 days
  The severity of coronary lesions is determined by using CAG/CTA and fractional flow reserve. Severe degree is defined as ≥90% stenosis of at least one main vessel or branch vessel with diameter ≥2mm. Moderate degree is defined as 50%-89% stenosis and fractional flow reserve ≤0.8. Mild degree is defined as <50% stenosis and fractional flow reserve ≤0.8, or stenosis 50%-89% and fractional flow reserve> 0.8. Sensitivity, specificity, and area under ROC curve (AUC) are performed for assessing the efficacy.
Efficacy of MCG in early stratification of patients with suspected NSTE-ACS | from the date of enrollment until the date of discharge, up to 30 days
  For early stratification measurement, patients with suspected NSTE-ACS are assessed by 30d (from enrollment) MACE and classified as high or low risk. Sensitivity, specificity, and area under ROC curve (AUC) are performed for assessing the efficacy of MCG.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguo Chen, Professor, Principal Investigator — Qliu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China